CLINICAL TRIAL: NCT04020237
Title: Evaluation of Quality of Life in Patients With Chronic Pulmonary Obstructive Disease According to Particular Matter Exposure
Brief Title: Impact of Particulate Matter in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sei Won Lee (Other)
Collaborators: Korea Centers for Disease Control & Prevention (Unknown)
Responsible Party: Sponsor-Investigator, Sei Won Lee, Clinical Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0476
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational arm (No Intervention): General counselling to particulate matter practice score.
- Interventional arm (Other): Active education and feedback on the particulate matter practice score that affects real life.
  Interventions: Behavioral: Education about particulate matter practice score

INTERVENTIONS:
Behavioral: Education about particulate matter practice score — For the intervention group, specific guidance is given to the patient who might be exposure in environment with higher particulate matter concentration.
  * 1) Start air purifier
  * 2) Do not go out and make it to the minimum when absolutely necessary
  * 3) It is recommended to wear a mask when going out.
  * 4) The investigators recommend a lot of water, fresh fruit and vegetables.
  * 5) Prepare an inhaler and use it when symptoms get worse.
  Arms: Interventional arm

SUMMARY:
A prospective study will be conducted in patients with COPD. The investigators will suggest about intervention for preventing in recurrence and aggravation of adult chronic respiratory disease due to exposure to particulate matter.

DETAILED DESCRIPTION:
Study trends and intervention plans related to particulate matter exposure and adult chronic respiratory disease in literature Measurement of particulate matter exposure by individual activities and collection of clinical information Linkage between individual particulate matter exposure and clinical information Investigation about effectiveness of intervention to avoid particulate matter

ELIGIBILITY:
Inclusion Criteria:

* COPD over 40 years of age
* Patients with pulmonary function tests with Forced expiratory volume at 1 second / forced vital capacity <0.7 and Forced expiratory volume at 1 second1 <80%

Exclusion Criteria:

* Patients under the age of 18
* Elderly people over 80 years old
* People with respiratory symptoms with modified Medical Research Council dyspnea scale 0
* Persons who do not understand the brief description of the particulate matter exposure device
* A person who does not agree to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-11 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Chage from life quality scale at 1 year | Up to 1 year
  Via average of total chronic obstructive pulmonary disease assessment test (CAT) score (total range 0-40, higher score means bad outcome, CAT score consisted of summed score about cough (0-5), phlegm (0-5), chest tightness (0-5), breathlessness (0-5), activites (0-5), confidence (0-5), sleep (0-5), energy (0-5))

SECONDARY OUTCOMES:
Change from pulmonary function test at 1 year | Up to 1 year
  Forced Expiratory Volume at 1 second level

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, Study Director — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Ra SW, Kang SY, Kim HC, Lee SW. Effect of particulate matter exposure on patients with COPD and risk reduction through behavioural interventions: the protocol of a prospective panel study. BMJ Open. 2020 Nov 9;10(11):e039394. doi: 10.1136/bmjopen-2020-039394. PMID 33168558